CLINICAL TRIAL: NCT01298505
Title: A Phase 1 Double-blind (3rd Party Open), Randomized, Placebo-controlled Study To Investigate The Safety And Toleration Of Multiple Oral Doses Of Pf-03654764 In Combination With Fexofenadine In Healthy Subjects
Brief Title: A Study To Investigate The Safety And Toleration Of Multiple Oral Doses Of PF-03654764 In Combination With Fexofenadine In Healthy Subjects
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: This study was stopped due to lack of evidence for clinical efficacy.
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: B0711006
Record Dates: First submitted 2011-02-02; First posted 2011-02-17 (Estimated); Last update posted 2019-02-11 (Actual); Status verified 2019-02

CONDITIONS: Healthy
Keywords: Phase 1 multiple dose safety toleration fexofenadine
MeSH Terms: interventions — 3-fluoro-3-(3-fluoro-4-(pyrrolidin-1-ylmethyl)phenyl)-N-(2-methylpropyl)cyclobutanecarboxamide; fexofenadine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- PF-03654764 2.5mg plus fexofenadine 60mg (Experimental)
  Interventions: Drug: PF-03654764 2.5mg plus fexofenadine 60mg
- PF-03654764 5mg plus fexofenadine 60mg (Experimental)
  Interventions: Drug: PF-03654764 5mg plus fexofenadine 60mg
- placebo (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: PF-03654764 2.5mg plus fexofenadine 60mg — PF-03654764 2.5mg plus fexofenadine 60mg twice daily for 7 days
  Arms: PF-03654764 2.5mg plus fexofenadine 60mg
Drug: PF-03654764 5mg plus fexofenadine 60mg — PF-03654764 5mg plus fexofenadine 60mg twice daily for 7 days
  Arms: PF-03654764 5mg plus fexofenadine 60mg
Drug: placebo — placebo given twice daily for 7 days
  Arms: placebo

SUMMARY:
The purpose of this study in heathy people is to investigate the safety, toleration and time course of PF-03654764 in the blood, following multiple doses given by mouth together with fexofenadine.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects. (Healthy is defined as no clinically relevant abnormalities identified by a detailed medical history, full physical examination, including blood pressure and pulse rate measurement, 12-lead ECG and clinical laboratory tests).

Exclusion Criteria:

* Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurologic, or allergic disease (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at time of dosing).
* A positive urine drug screen.
* Treatment with an investigational drug within 30 days (or as determined by the local requirement, whichever is longer) or 5 half-lives preceding the first dose of study medication.

Ages: 21 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2010-06-04 (Actual); Primary Completion 2010-06-04 (Actual); Study Completion 2010-06-04 (Actual)

PRIMARY OUTCOMES:
Number of participants with adverse events as a measure of safety and tolerability. | 30 days

SECONDARY OUTCOMES:
Plasma concentrations of PF-03654764 will be measured. | 7 days

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Clinical Research Unit, Singapore, Singapore

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B0711006&StudyName=A%20Study%20To%20Investigate%20The%20Safety%20And%20Toleration%20Of%20Multiple%20Oral%20Doses%20Of%20PF-03654764%20In%20Combination%20With%20Fexofenadine%20In%20Healthy%20Sub